CLINICAL TRIAL: NCT04005833
Title: Association Between Blood Fibrocytes During an Exacerbation and Lung Function Decline in Patients With Early Stage Chronic Obstructive Pulmonary Disease (COPD) in Primary Care
Brief Title: Blood Fibrocytes During an Exacerbation and Lung Function Decline in Patients With COPD in Primary Care.
Acronym: FIBRO-COPD
Status: Terminated | Type: Observational
Why Stopped: Inclusions were suspended due to the COVID-19 pandemic, and the inclusion rate would not increase during the resumption.
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2017/43
Record Dates: First submitted 2019-02-15; First posted 2019-07-02 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary disease; chronic obstructive; Primary Health Care; Fibrocyte; Respiratory Function Tests
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Specific to research: the determination of fibrocytes on EDTA tubes (with Ethylenediaminetetraacetic acid) The samples will be transported fresh to measure the rate of circulating blood fibrocytes by flow cytometry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD exacerbation: COPD exacerbation, compared according to blood fibrocytes level measured during the suspected exacerbation (Day 1)
  Interventions: Diagnostic Test: spirometry

INTERVENTIONS:
Diagnostic Test: spirometry — The lung function (FEV1) will be assessed at follow-up visits at 2 months, 12 months and 36 months after inclusion.

SUMMARY:
This study aims to estimate the association between blood fibrocytes measured during a suspected exacerbation and 3-year decline forced expiratory volume in one second (FEV1), in patients with Chronic obstructive pulmonary disease (COPD) in primary care, with a history of smoking, independently of the number of exacerbations and of tobacco or occupational exposure.

DETAILED DESCRIPTION:
COPD is highly prevalent in primary care. It is associated with tobacco smoke or toxic occupational exposure. Some COPD patients will experience a faster decline in quality of life and lung function. There is currently no prognostic marker allowing to identify those patients at higher risk of fast lung function decline. Recent data suggest that fibrocytes are involved in COPD's physiopathology. A higher blood fibrocytes level during an acute exacerbation has been associated with higher mortality in COPD patients at a late stage of the disease. In mice, fibrocytes role in lung function decline has been demonstrated at an early stage. To date, association between blood fibrocytes during an exacerbation and lung function decline has not been evaluated at the early stage of COPD in humans.

This study aims to estimate the association between blood fibrocytes measured during a suspected exacerbation and 3-year decline in forced expiratory volume in one second (FEV1), in patients with COPD in primary care, with a history of smoking, independently of the number of exacerbations and of tobacco or occupational exposure.

In this study, blood fibrocytes during a suspected exacerbation will be measured at inclusion. The lung function (FEV1) will be assessed at follow-up visits at 2 months, 12 months and 36 months after inclusion. COPD-related health status and severity of dyspnea will be assessed with COPD Assessment test (CAT) and the modified Medical Research Council dyspnea scale (mMRC) at follow-up visits at 2 months, 12 months and 36 months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* man or woman aged more than 40 years old,
* with tobacco exposure of more than 20 pack-years,
* Presenting to a General Practitioner with a suspected mild or moderate COPD exacerbation according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines (worsening of symptoms with the need for prescribing short acting bronchodilatators, antibiotics or oral corticosteroids)
* Informed consent given
* Affiliated to a social insurance scheme

Exclusion Criteria:

* Severe exacerbation of COPD according to GOLD guidelines (patient requires hospitalization or visits to the emergency room),
* More likely differential diagnosis than a COPD exacerbation, such as pneumonia, acute pulmonary oedema or other differential diagnosis,
* history of asthma, pulmonary fibrosis, primary pulmonary hypertension or chronic viral infections (HIV, hepatitis)
* person under care or protection of vulnerable adults

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Man or woman aged more than 40 years old with tobacco exposure of more than 20 pack-years, Presenting to a General Practitioner with a suspected mild or moderate COPD exacerbation according to GOLD guidelines (worsening of symptoms with the need for prescribing short acting bronchodilatators, antibiotics or oral corticosteroids).
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
number of blood fibrocytes | Day 1
  blood fibrocytes level measured during the suspected exacerbation
Forced Expiratory Volume (FEV) | month 36
  FEV1 assessed by spirometry

SECONDARY OUTCOMES:
Forced Expiratory Volume (FEV) | month 2
  FEV1 assessed by spirometry
Forced Expiratory Volume (FEV) | month 12
  FEV1 assessed by spirometry
Score of modified Medical Research Council dyspnea scale | month 2
  The MMRC dyspnea scale is a standardized questionnaire validated and measuring the degree of dyspnea in patients with COPD. The scale is an ordinal variable into 5 classes from 0 to 4, a score of 4 representing a major dyspnea.
Score of modified Medical Research Council dyspnea scale | month 12
  The MMRC dyspnea scale is a standardized questionnaire validated and measuring the degree of dyspnea in patients with COPD. The scale is an ordinal variable into 5 classes from 0 to 4, a score of 4 representing a major dyspnea.
Score of modified Medical Research Council dyspnea scale | month 36
  The MMRC dyspnea scale is a standardized questionnaire validated and measuring the degree of dyspnea in patients with COPD. The scale is an ordinal variable into 5 classes from 0 to 4, a score of 4 representing a major dyspnea.
Score of Chronic obstructive pulmonary disease Assessment Test | month 2
  health status measured by CAT (http://www.catestonline.org/english/index_France.htm)
Score of Chronic obstructive pulmonary disease Assessment Test | month 12
  health status measured by CAT (http://www.catestonline.org/english/index_France.htm)
Score of Chronic obstructive pulmonary disease Assessment Test | month 36
  health status measured by CAT (http://www.catestonline.org/english/index_France.htm)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Prothon, MD, Principal Investigator — University of Bordeaux; Patrick Berger, MD/PhD, Study Chair — Hospital University, Bordeaux
Locations (2):
- France (2):
  - Cabinet médical, Belin-Béliet
  - Cabinet Médical, Cadillac

IPD SHARING:
Plan to Share IPD: No